CLINICAL TRIAL: NCT04310397
Title: Altering Adjuvant Therapy Based on Pathologic Response to Neoadjuvant Dabrafenib and Trametinib (ALTER-PATH NeoDT)
Brief Title: Dabrafenib, Trametinib, and Spartalizumab for the Treatment of BRAF V600E or V600K Mutation Positive Stage IIIB/C/D Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to slow enrollment
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0906; NCI-2020-00941 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0906 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-03-04; First posted 2020-03-17 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8
Keywords: Melanoma; Neoadjuvant; Pathological Response; Targeted Therapy; Immunotherapy
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; spartalizumab; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dabrafenib, trametinib, surgery, spartalizumab) (Experimental): NEOADJUVANT TREATMENT: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28. Treatment repeats every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  SURGERY: Patients undergo surgical resection of melanoma.
  ADJUVANT TREATMENT OF pCR PATIENTS: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28. Cycles repeats every 28 days for 44 weeks in the absence of disease progression or unacceptable toxicity.
  ADJUVANT TREATMENT OF NON pCR PATIENTS: Patients receive spartalizumab IV over 30 minutes on day 1, dabrafenib PO BID and trametinib PO QD on days 1-28. Cycles repeats every 28 days for 44 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dabrafenib; Biological: Spartalizumab; Procedure: Therapeutic Conventional Surgery; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Given PO
  Other Names: BRAF Inhibitor GSK2118436; GSK-2118436; GSK-2118436A; GSK2118436
Biological: Spartalizumab — Given IV
  Other Names: PDR-001; PDR001
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
This phase II trial studies how well dabrafenib, trametinib, and spartalizumab works in treating patients with BRAF V600E or V600K mutation positive stage IIIB/C/D melanoma, who do not achieve a pathologic complete response after 8 weeks of dabrafenib and trametinib treatment. Patients who achieve a pathologic complete response after 8 weeks of neoadjuvant dabrafenib and trametinib will receive adjuvant dabrafenib and trametinib. Dabrafenib and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as spartalizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving dabrafenib, trametinib, and spartalizumab may help to control melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the 12-month relapse free survival (RFS) rate in stage IIIB/C/D melanoma patients who, after 8 weeks of neoadjuvant dabrafenib and trametinib, do not achieve a pathologic complete response (pCR) and receive adjuvant dabrafenib, trametinib and spartalizumab.

SECONDARY OBJECTIVES:

I. To evaluate the safety of neoadjuvant dabrafenib and trametinib and adjuvant dabrafenib, trametinib and spartalizumab.

II. To determine the 12-month relapse free survival (RFS) rate in stage IIIB/C/D.

III. Melanoma patients who, after 8 weeks of neoadjuvant dabrafenib and trametinib, achieve a pCR and receive adjuvant dabrafenib and trametinib.

IV. To assess the recurrence patterns, distant metastasis-free survival (DMFS), and overall survival (OS) in all patients treated on protocol.

EXPLORATORY OBJECTIVES:

I. To assess immunological and molecular features of treatment response and resistance.

II. To assess circulating markers and correlate them with treatment response and relapse and toxicity III. To assess the impact of neoadjuvant therapy on surgical resectability.

OUTLINE:

NEOADJUVANT TREATMENT: Patients receive dabrafenib orally (PO) twice daily (BID) and trametinib PO once daily (QD) on days 1-28. Treatment repeats every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity.

SURGERY: Patients undergo surgical resection of melanoma.

ADJUVANT TREATMENT OF pCR PATIENTS: Patients receive dabrafenib PO BID and trametinib PO QD on days 1-28. Cycles repeats every 28 days for 44 weeks in the absence of disease progression or unacceptable toxicity.

ADJUVANT TREATMENT OF NON pCR PATIENTS: Patients receive spartalizumab intravenously (IV) over 30 minutes on day 1, dabrafenib PO BID and trametinib PO QD on days 1-28. Cycles repeats every 28 days for 44 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-4 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Patients must have histologically or cytologically confirmed clinically detected, node involved Stage IIIB/C/D melanoma by American Joint Committee on Cancer (AJCC) version 8 and surgically resectable disease. The definition of resectability can be determined by the patient's surgical oncologist and verified via discussion at multidisciplinary tumor conference attended by melanoma medical and surgical oncology staff. Resectable tumors are defined as having no significant vascular, neural or bony involvement that would preclude complete resection or necessitate the use of adjuvant radiation. Only cases where a complete surgical resection with tumor- free margins can safely be achieved are defined as resectable
* BRAF mutation-positive melanoma (V600E or V600K) based on report from a Clinical Laboratory Improvement Act (CLIA) certified laboratory
* Patients must have measurable disease, defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Patients who have been previously treated in the adjuvant setting with ipilimumab or interferon alpha or investigational vaccines for melanoma will be eligible for treatment after a 28 day wash-out period
* Patients who have previously received anti PD-1 in the adjuvant setting will be allowed if it has been six months or longer since previous drug exposure
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant will be required to use highly effective methods of contraception during dosing and for 150-days after stopping treatment with spartalizumab. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject
  * Placement of a non-hormonal intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
  * Notes:

    * Double-barrier contraception: condom and occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/cream/suppository) are not considered highly effective methods of contraception.
    * Hormonal-based methods (e.g., oral contraceptives) are not considered as highly effective methods of contraception due to potential drug-drug interactions with dabrafenib.
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential
* Sexually active males must use a condom during intercourse while on treatment and for 150 days after stopping treatment with spartalizumab and should not father a child in this period. A condom is required to be used by vasectomized men as well during intercourse in order to prevent delivery of the drug via semen
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x ULN
* International normalized ratio (INR) OR prothrombin time (PT) =<1.5 x ULN unless participant is receiving anticoagulant therapy as long as prothrombin time (PT) or partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug within 28 days
* Evidence of metastatic melanoma or patients with only in-transit metastases without involved nodes
* Prior BRAF or MEK inhibitor use
* Prior anti PD-1 or anti PD-L1 inhibitor use in last 6 months
* Prior malignancy active within the previous 2 years except for patient's prior diagnosis of melanoma and locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast with local control measures (surgery, radiation)
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Any positive test result for hepatitis B or C and human immunodeficiency virus (HIV) virus indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome
* History of severe hypersensitivity reaction to any monoclonal antibody
* History of Central serous retinopathy (CSR) or retinal vein occlusion (RVO), or predisposing factors to RVO or CSR (e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs
* Corrected QT (QTc) interval >= 480 msec (>= 500 msec for subjects with bundle branch block)
* Uncontrolled arrhythmias
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
* Pregnant or lactating female
* Unwillingness or inability to follow the procedures required in the protocol
* Uncontrolled diabetes, hypertension or other medical conditions that may interfere with assessment of toxicity
* Subjects with known glucose 6 phosphate dehydrogenase (G6PD) deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N Amaria, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with resectable stage IIIB/IIIC/IIID melanoma with BRAF V600E/K mutations. Only patients with V600E or V600K mutations are eligible for enrollment. Patients with BRAF by IHC is acceptable to for screening.
Pre-assignment Details: 4 patients consented and treated.
Groups:
- Arm 1: Dabrafenib 150 mg PO BID D1-28 (starting dose); trametinib PO QD D1-28 (starting dose); Spartalizumab 400 mg IV over 30 minutes every 28 days
Period: Overall Study
Arm/Group | Arm 1
Started | 4
Completed | 0
Not Completed | 4
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate in Stage IIIb/C/D Subjects
Description: To determine the 12-month relapse free survival (RFS) rate in stage IIIB/C/D melanoma patients who, after 8 weeks of neoadjuvant dabrafenib and trametinib, do not achieve a pCR and receive adjuvant dabrafenib, trametinib an spartalizumab.
Time Frame: Baseline up to 2 years
Population: Data were not collected
Arm/Group | Arm 1
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety of Neoadjuvant Treatments
Description: To evaluate the sarety of neoadjuvant dabrafenib and trametini and adjuvant dabrafenib, trametinib ann spartalizumab
Time Frame: Baseline up to 2 years
Population: Data were not collected
Arm/Group | Arm 1
Number analyzed (Participants) | 0

3. Secondary Outcome: Distant Metastasis-free Survival (DMFS) and Overall Survival (OS)
Description: To assess the recurrence patterns, distant metastasis-free survival (DMFS), and overall survival (OS) in all patients treated on protocol.
Time Frame: Baseline upto 2 years
Population: Data were not collected
Arm/Group | Arm 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 2 years
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=4)
Fever (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Soft Tissue Infection (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransfease increased (Investigations) | 3 (8)
Alkaline amionotransferase (Investigations) | 3 (5)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 3 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Elevated WBC (Blood and lymphatic system disorders) | 2 (2)
Increased ANC (Blood and lymphatic system disorders) | 2 (2)
Blurred Vision (Eye disorders) | 1 (1)
Chills (General disorders) | 4 (16)
Constipation (Gastrointestinal disorders) | 3 (4)
Creatinine Increased (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT04310397/Prot_SAP_000.pdf